CLINICAL TRIAL: NCT00328575
Title: Phase I Dose Escalation Trial in Patients With Brain Metastases Using IMRT
Brief Title: Using Intensity Modulated Radiation Therapy (IMRT) for Brain Metastases
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sidney Kimmel Cancer Center at Thomas Jefferson University (Other)
Responsible Party: Sponsor
Organization: Thomas Jefferson University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 05U.443; 2005-70 (Other: CCRRC); 05U.443R (Other: IRB)
Record Dates: First submitted 2006-05-19; First posted 2006-05-22 (Estimated); Last update posted 2016-10-21 (Estimated); Status verified 2016-10

CONDITIONS: Neoplasm Metastasis
Keywords: Brain metastases; Parenchymal; Neoplasm; IMRT; Intensity Modulated Radiation Therapy
MeSH Terms: conditions — Neoplasm Metastasis; Brain Neoplasms; Neoplasms | interventions — Radiotherapy, Intensity-Modulated; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Intensity-Modulated Radiotherapy (IMRT) (Experimental): Patients with brain metastases will be enrolled in one of three dose levels based on tumor size. For tumor size of 3 cm or less (maximum diameter in any dimension), doses of 47.5Gy, 52.5Gy, and 54.5Gy will be tested. For tumor size of greater than 3 cm (maximum diameter in any dimension), doses of 42.5Gy, 47.5Gy, and 52.5Gy will be tested.
  Interventions: Radiation: Intensity-Modulated Radiotherapy (IMRT)

INTERVENTIONS:
Radiation: Intensity-Modulated Radiotherapy (IMRT) — The duration of radiation therapy will be total of 3 weeks. During the first week, all patients will be treated initially with whole brain radiation therapy (WBRT) at 2.5Gy per fraction daily 5 days a week to a dose of 12.5Gy. This will be delivered through parallel-opposed fields to cover the entire cranial contents.
  For the remaining 2 weeks, patients will be treated using intensity-modulated radiation therapy (IMRT) technology such that a higher dose can be delivered to the tumor. IMRT is capable of generating complex 3-D dose distribution to conform closely to the target volume by modulating the radiation beam. This process is based on the "inverse method" of treatment planning to optimize radiation dose to tumor target coverage and normal tissue sparing.
  Other Names: Radiation Therapy

SUMMARY:
The purpose of this study is to determine if using intensity modulated radiation therapy for brain metastases is safe and will improve local control more than standard whole brain radiation therapy.

DETAILED DESCRIPTION:
Traditionally, whole brain radiation therapy (WBRT) has been the primary therapy for patients with brain metastases. Despite this therapy, patients still have poor survival of four to six months. Untreated patients have a median survival of one month. Up to one half of these patients die of causes related to the presence of brain metastases. In a Phase I/II RTOG trial, the efficacy and safety of delivering accelerated fractionation was investigated in patients with good prognostic factors. No toxicity was observed with escalating dose of irradiation up 70.40Gy in 1.6Gy twice daily treatments. However, in a randomized trial, the use of hyperfractionation did not appear to improve survival when compared to 30Gy whole brain irradiation delivered in 10 fractions.

Current therapeutic approach also includes stereotactic radiosurgery (SRS). Several retrospective studies have demonstrated improved local tumor control of 80% with addition of SRS to WBRT. These local control rates were comparable to surgery. In a recently published randomized trial by RTOG 95-08 (TJU accrued 42 patients to this trial), Andrews et al. demonstrated improved survival in patients with solitary brain lesion treated with SRS. Median survival was 6.5 months in patients treated with WBRT and SRS compared to 4.9 months in patients treated with WBRT alone. Also, these patients were more likely to have stable or improved performance status.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed malignancy
* 2-5 parenchymal brain metastases on magnetic resonance imaging (MRI) with a maximum size of 4 cm
* Partial resection allowed. Complete resection allowed only in patients with more than 3 lesions.
* Karnofsky Performance Status (KPS) equal to or greater than 60
* Neurologic function equal to or greater than 2

Exclusion Criteria:

* Recurrent brain tumors
* Major medical or psychiatric illnesses
* Metastases in brainstem, midbrain, pons, or medulla
* Patients with leukemia or lymphoma

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2005-10; Primary Completion 2009-07 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Unacceptable Acute CNS Toxicity | 3 weeks
  The primary endpoint is the frequency of patients developing unacceptable acute CNS toxicity.

SECONDARY OUTCOMES:
Dose-Limiting Toxicity (DLT) | 30 days
  Dose-limiting toxicity will be defined as Grade 3 or greater CNS toxicity, as per NCI criteria. The observed rate of > 30% of Grade 3 or greater acute CNS toxicities will be considered unacceptable. Late toxicities will be closely monitored as well.

CONTACTS AND LOCATIONS:
Overall Officials: Wenyin Shi, MD, PhD, Principal Investigator — Thomas Jefferson University
Locations (1):
- Thomas Jefferson University, Philadelphia, Pennsylvania, United States

REFERENCES:
- See also: Kimmel Cancer Center at Thomas Jefferson University, an NCI-Designated Cancer Center — http://www.KimmelCancerCenter.org